CLINICAL TRIAL: NCT05320874
Title: The Safety, Tolerability, Pharmacokinetic Characteristics and Efficacy of KM257 in Patients With Advanced HER2-positive or Expressing Solid Tumors in a Single-arm, Open-label, Multi-center Phase 1 Clinical Study.
Brief Title: A Study of KM257 in Patients With Advanced HER2-positive or Expressing Solid Tumors.
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xuanzhu Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KM257-1001
Record Dates: First submitted 2022-04-01; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Advanced Solid Tumor
Keywords: KM257; Safety, tolerability, pharmacokinetics and efficacy; Advanced HER2 positive or expressing solid tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KM257 (Experimental): KM257 Bispecific antibody
  Interventions: Biological: KM257 Bispecific antibody

INTERVENTIONS:
Biological: KM257 Bispecific antibody — Part 1a dose escalation:
  There will be 3 increasing dose levels (3mg/kg,6mg/kg,12mg/kg). Patients will be intravenously administrated with one dose of KM257, QW for continuous cycles of 21 consecutive days for each cycle. The dosing interval may be adjusted during the study based on emerging data from this trial.
  Part 1b dose expansion:
  Part1b:For cohort 1 and cohort2, KM257 will be given at the RP2D identified in Part1a;
  For cohort 3 to 7:KM257 will be given combined with one of the following selected drug combination:
  Drug: Capecitabine Combination therapy with KM257 - Cohort 3
  Drug: Paclitaxel or Docetaxel or Irinotecan Combination therapy with KM257 - Cohort 4
  Drug: Gemcitabine+Cisplatin Combination therapy with KM257 - Cohort 5
  Drug: Gemcitabine+Cisplatin or Carboplatin Combination therapy with KM257 - Cohort 6
  Drug:Carboplatin+Paclitaxel Combination therapy with KM257 - Cohort 7

SUMMARY:
This is a first-in-human, 2-part study to investigate the safety, tolerability, pharmacokinetics and efficacy of KM257 by itself and combined with selected chemotherapy agents in patients with advanced HER2-positive or expressing cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand, voluntarily participate and willing to sign the ICF.
2. Male or female subject >= 18 years and =<75 years.
3. Histologically or cytologically confirmed advanced solid tumors.
4. HER2 positive or expressing.
5. ECOG score 0 or 1.
6. According to the definition of RECIST1.1, for Part1a, the patient has evaluable but Non-measurable lesion can be accepted. For Part1b, the patient has at least one measurable lesion.
7. Life expectancy≥12weeks.
8. Adequate organ function.
9. Subjects (women of child-bearing potential and males with fertile female partner) must be willing to use viable contraception method.

Exclusion Criteria:

1. primary CNS tumors (including meningeal tumors), symptomatic or untreated CNS metastases(including meningeal metastases).
2. Subjects who had other malignancies in the 2 years prior to the first administration of the investigational drug were excluded in Phase Ib, except those who had basal cell carcinoma, breast cancer in situ, or cervical cancer in situ and had no recurrence and metastasis after radical therapy.
3. Accepted any other anti-tumor drug therapies within 2 weeks before first dose.
4. Accepted major surgery or radical radiotherapy within 4 weeks before first dose; Accepted palliative radiotherapy within 2 weeks before first dose; Accepted radioactive agents(strontium, samarium, etc.)for therapeutic purposes within 8 weeks before first dose.
5. Participating in other studies involving investigational drug(s) ≤ 4 weeks before the first dose of KM257.
6. Subjects with interstitial lung disease or non-infectious pneumonia and related history.
7. Infection with HIV disease.
8. Active hepatitis.
9. Had an active infection requiring systemic treatment within 2 weeks prior to initial administration of the investigational drug.
10. Cavity effusion (pleural effusion, ascites, pericardial effusion, etc.) are not well controlled.

    Subjects are eligible with clinically controlled and stable neurologic function >= 4 weeks, which is no evidence of CNS disease progression; Subjects with
11. Subjects who have received organ transplants.
12. Unresolved toxicities ( Common Terminology Criteria for Adverse Event (CTCAE, version 5), grade greater than or equal to2) from prior anti-cancer therapy. (with the exception of alopecia, the special provisions of inclusion criteria);
13. Subjects who have a history of severe allergic reactions to antibody medications or have a history of severe allergic asthma (CTCAE V5.0 grade ≥3).
14. Subjects with a known history of alcohol or drug abuse.
15. History of myocardial infarction or unstable angina within 6 months prior to enrollment, congestive heart failure (NYHA Class≥2), or clinically significant cardiac disease，LVEF<50%，QTc Fridericia (QTcF) > 470 ms for female, QTc Fridericia (QTcF) > 450 ms for male.
16. History of TIA or stroke within 6 months prior to initial administration of KM257.
17. Subjects known to have a mental illness that may affect trial compliance.
18. The investigator considers that the subject has any clinical or laboratory abnormalities or other reasons that would disqualify him or her from participating in this clinical study.
19. Part1b cohort 2: subjects with known mutations in exons 2, 3, and 4 of KRAS/NRAS and in V600E of BRAF.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) (Part 1a) | Up to 3 weeks
  Determine maximum tolerated dose (MTD) of KM257.
Recommended phase 2 dose (RP2D) (if has) (Part 1a) | Up to 3 weeks
  Determine recommended phase 2 dose (RP2D) of KM257.
Number of patients with adverse events.(Part 1a) | Up to 8 months.
  Number of patients who experienced an adverse event
Objective response rate (ORR) (Part 1b) | Up to 2-3 years.
  Number of participants who achieved a best response of either complete response (CR) or partial response (PR) during treatment evaluated by investigators according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Area under the concentration versus time curve of KM257 in plasma (AUC) (Part 1a and Part1b). | Up to 8 months for Part 1a; Up to 2 to 3 years for Part1b.
  To determine the AUC of KM257.
Maximum serum concentration (Cmax) of KM257(Part 1a and Part 1b ). | Up to 63days for Part 1a; Up to 63 days for Part1b.
  To determine the maximum serum concentration (Cmax) of KM257.
Time of Maximum observed serum concentration (Tmax) of KM257 (Part1 and Part1b ) . | Up to 63days for Part 1a; Up to 63days for Part1b.
  To determine the Tmax of KM257.
Serum Half-life (T-HALF) of KM257. (Part1a and Part1b) | Up to 63days.
  To determine the t1/2 of KM257.
Frequency and titer of anti-KM257 antibody. (Part1a and Part1b) | up to 8months for Part1a and up to 2-3 years for Part1b.
  To determine the immunogenicity of KM257.
Objective response rate (ORR) (Part 1a) | Up to 8months.
  Number of participants who achieved a best response of either complete response (CR) or partial response (PR) during treatment evaluated by investigators according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Progression free survival (PFS) (Part 1a and Part 1b) | up to 2-3 years.
  To determine the PFS by investigator.
Disease control rate (DCR) (Part 1a and Part 1b) | up to 2-3 years.
  To determine the DCR by investigator.
Overall survival (OS) (Part1a and Part1b ) | up to 2-3 years.
  To determine the OS by investigator.
Number of patients with adverse events (Phase 1b) | up to 2-3 years.
  Incidence of AE as assessed by CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China